CLINICAL TRIAL: NCT05358080
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Superiority, Phase IV Trial to Evaluate the Efficacy and Safety of Entelon 50mg Compared to Placebo in Patients With Non-Proliferative Diabetic Retinopathy
Brief Title: Study to Evaluate Efficacy and Safety of Entelon 50mg in Patients With Non-Proliferative Diabetic Retinopathy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HL-ENTL-402
Record Dates: First submitted 2022-04-25; First posted 2022-05-03 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Non Proliferative Diabetic Retinopathy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Entelon Tab. 50mg (Experimental)
  Interventions: Drug: Entelon Tab. 50mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Entelon Tab. 50mg — twice daily for 24months
  Other Names: Vitis Vinifera Seed Dreid Extract 50mg
  Arms: Entelon Tab. 50mg
Drug: Placebo — twice daily for 24months
  Arms: Placebo

SUMMARY:
This clinical trial is a multi-center, double-blind, randomized, placebo controlled , parallel design, superiority, phase 4 study to evaluate the efficacy and safety of Entelon 50mg in 396 patients with non-proliferative diabetic retinopathy.

DETAILED DESCRIPTION:
This study is to prove that Entelon tab. 50mg is superior in clinical efficacy and safety compared to placebo for 24 months in patients suffering from non-proliferative diabetic retinopathy.

ELIGIBILITY:
Inclusion Criteria:

1. 19 years ≤ age
2. Those who are diagnosed as Type 2 diabetes mellitus
3. Those whose blood sugar level has been well adjusted to less than 9% of HbA1c with dietary and oral blood sugar lowering durgs for 3 months based on the time of screening
4. Those who agree to use an effective method of contraception
5. Those who provide written consent voluntarily to participate in this clinical trial

Inclusion criteria for the study eye

1. Those with 0.5(20/40 Snellen lines) or more visual acuity
2. Those with 300 micrometers or less central macular thickness
3. Those who are diagnosed as mild to moderate NPDR(DRSS levels 35-47)

Exclusion Criteria:

1. Those who are diagnosed as proliferative diabetic retinopathy
2. Those with macular edema
3. Diabetic subjects who have difficulty in controlling blood sugar
4. Those whose blood pressure is not well controlled at the time of the screening(>140/90mmHg)
5. Those who, have had stroke or myocardial infarction or arrhythmia that should be treated within 6 months prior to the time of screening
6. Subjects with severe renal disorder or severe liver disorder
7. Those who have a history of malignant tumors within 5 years prior to the time of screening
8. Those who are required to receive Kallidinogenase, Vaccinium myrtillus extract, Sulodexide, or Calcium dobesilate during the clinical trial period
9. Those who have an allergy to investigational product or any of its excipients
10. Those who have an allergy to fluorescein
11. Those who have galactose intolerance, lapp lactase deficiency, or glucose-galactose malabsorption
12. Those who have difficulty to get OCT test or Fundus photo test
13. Pregnant or lactating woman
14. Those with medication of other investigational product within 3 months prior to the time of randomization
15. Patients who are considered to be ineligible for study participation by the investigator

Exclusion criteria for the study eye

1. Those who have a visual defect that can affect the evaluation determined by an investigator
2. Those who have a opacity that can affect the evaluation determined by an investigator
3. Those who have eye diseases that can affect the evaluation determined by an investigator
4. Those with 25mmHg or more intraocular pressure on a study eye
5. Those who are on medication of intravitreal injection of steroid or anti VEGF treatment or get laser photocoagulation within 6 months prior to the first administration
6. Those who have a history of a vitrectomy
7. Those who have a major ophthalmic surgery history within 3 months prior to the time of first administration for investigational products
8. Those who have a history of yttrium aluminum garnet capsulotomy within 2 months prior to the time of first administration for investigational products
9. Those with a phakia

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Estimated)
Dates: Start 2022-05-27 (Actual); Primary Completion 2024-12-16 (Estimated); Study Completion 2024-12-16 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects maintained or improved in DRSS level | 24 months(Visit 10)
  Change at 24 months of treatment with the drug from baseline(day 0) in DRSS(Diabetic Retinopathy Severity Scale) level

SECONDARY OUTCOMES:
Proportion of subjects maintained or improved in DRSS level | 12 months(Visit 6)
  Change at 12 months of treatment with the drug from baseline(day 0) in DRSS(Diabetic Retinopathy Severity Scale) level
Proportion of subjects maintained or improved or worsened in DRSS | 12 months(Visit 6), 24 months(Visit 10)
  Percentage of subjects with no change in DRSS(diabetic retinopathy severity scale) compared to baseline at 12 or 24 months compared to baseline, improved one or more levels, improved two or more levels, worsened one or more levels, and worsened two or more levels
Amount of change BCVA letter | 24 months(Visit 10)
  Amount of change in BCVA(best corrected visual acuity) letters at 24 months relative to baseline
Proportion of subjects improved or worsened in BCVA | 24 months(Visit 10)
  Proportion of subjects with improved five or more letters in BCVA(best corrected visual acuity) and worsened five or more letters at 24 months compared to baseline
Change in quantitative of hard exudate | 6 months(Visit 4), 12 months(Visit 6), 18 months(Visit 8), 24 months(Visit 10)
  Amount and rate of change in quantitative of hard exudate through fundus photo
Change in CMT and TMV | 6 month(Visit 4), 12 month(Visit 6), 18 month(Visit 8), 24 month(Visit 10)
  Amount of change in CMT(Central macular thickness) and TMV(Total macular volume)
Proportion of subjects with CSME | through study completion, an average of 2 years
  Proportion of subjects with CSME(Clinically significant macular edema)

CONTACTS AND LOCATIONS:
Overall Officials: Ha Kyoung Kim, Principal Investigator — Hallym University Kangnam Sacred Heart Hospital
Locations (1):
- Hallym University Kangnam Sacred Heart Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No